CLINICAL TRIAL: NCT03401450
Title: Optimal Location of Nerve Block to Minimize Perioperative Opioid Administration in ACL Surgery: Comparing True Adductor Canal to Proximal Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-01602
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Results first posted 2020-12-23 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: ACL Surgery
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACB within true AC with bupivacaine (Active Comparator): The patients will receive an ultrasound-guided single injection adductor canal block with 20 mL of 0.5% bupivacaine
  Interventions: Drug: ACB within true AC with bupivacaine 0.5% 20cc
- ACB proximal to true AC with bupivacaine (Active Comparator): The patients will receive an ultrasound-guided single injection femoral triangle block with 20 mL of 0.5% bupivacaine
  Interventions: Drug: ACB proximal to true AC with bupivacaine 0.5% 20cc

INTERVENTIONS:
Drug: ACB within true AC with bupivacaine 0.5% 20cc — The adductor canal block (ACB) is more commonly being used to provide post-operative analgesia since it provides a sensory block with minimal motor block.
  Other Names: bupivacaine
  Arms: ACB within true AC with bupivacaine
Drug: ACB proximal to true AC with bupivacaine 0.5% 20cc — Patients will receive ultra-sound guided single femoral triangle block injection with 20 mL of 0.5% bupivicaine
  Other Names: bupivacaine
  Arms: ACB proximal to true AC with bupivacaine

SUMMARY:
This is a prospective, randomized, single blinded trial involving human subjects. The goal of this study is to determine an optimal location (proximal or distal) for the nerve block and whether it will make a difference in how much opioid the patient will receive during and after surgery. Ultrasound will identify the adductor canal and the proximal end of the adductor canal/apex of the femoral triangle to determine the location of the blocks.

Their will be two randomized groups: 1. ACB within true AC with bupivacaine 0.5% 20cc2. ACB proximal to true AC with bupivacaine 0.5% 20cc

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral, ACL surgery with allograft.
* Patients who consent to be randomized.
* Patients must be English proficient.

Exclusion Criteria:

* Patients younger than 18 or older than 75 years of age;
* Patients with a history of chronic pain or who are taking medications intended to treat chronic pain such as strong opioids;
* Patients with history of neurologic disorder that can interfere with pain sensation;
* Patients with a history of drug or alcohol abuse;
* Patients who are unable to understand or follow instructions;
* Patients with an allergy or a contraindication to any of the medications used in the study, or patients with a contraindication to any of the study procedures;
* Patients with severe liver disease, renal insufficiency, congestive heart failure, and/ or significant heart disease;
* Patients with a BMI over 42;
* Any patient that the investigators feel cannot comply with all study related procedures.
* Patients who do not tolerate Percocet.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prianka Desai, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACB Within True AC With Bupivacaine | ACB Proximal to True AC With Bupivacaine
Started | 33 | 36
Completed | 21 | 23
Not Completed | 12 | 13
Not completed — Lost to Follow-up | 4 | 6
Not completed — Anesthesia plan changed | 2 | 2
Not completed — Did not complete medication diary | 4 | 2
Not completed — post surgery medication change | 2 | 1
Not completed — Cancelled surgery | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACB Within True AC With Bupivacaine | ACB Proximal to True AC With Bupivacaine | Total
Number analyzed (Participants) | 33 | 36 | 69
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 10 | 9 | 19
  26-35 years | 13 | 15 | 28
  36-45 years | 3 | 7 | 10
  46-55 years | 6 | 5 | 11
  56-65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 19 | 19 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 23 | 21 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 33 | 36 | 69

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption Intraop Measured by Amounts of Morphine Equivalents
Description: Amount of morphine equivalents administered intraoperatively in 24 hours
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: milligrams of morphine equivalents
Arm/Group | ACB Within True AC With Bupivacaine | ACB Proximal to True AC With Bupivacaine
Number analyzed (Participants) | 21 | 23
milligrams of morphine equivalents | 23.21 (12.23) | 18.93 (9.34)

2. Primary Outcome: Total Opioid Consumption Postop Measured by Amounts of Morphine Equivalents
Description: Amount of morphine equivalents administered postoperatively in 24 hours
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: mg of morphine equivalents
Arm/Group | ACB Within True AC With Bupivacaine | ACB Proximal to True AC With Bupivacaine
Number analyzed (Participants) | 21 | 23
mg of morphine equivalents | 10 (6.79) | 13.18 (7.57)

3. Primary Outcome: Side Effects Such as Nausea, Itching, Constipation.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | ACB Within True AC With Bupivacaine | ACB Proximal to True AC With Bupivacaine
Number analyzed (Participants) | 21 | 23
Participants | 0 | 0

4. Secondary Outcome: Motor Block (Muscle Weakness): in PACU and Measured in Surgeons' Clinic at 3, 6 and 12 Months.
Time Frame: 12 months
Population: This measure was not measured/assessed in study participants; the orthopedic surgeon's office did not perform this test in the clinic at any point of the study.
Arm/Group | ACB Within True AC With Bupivacaine | ACB Proximal to True AC With Bupivacaine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | ACB Within True AC With Bupivacaine | ACB Proximal to True AC With Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 0/20 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT03401450/Prot_SAP_000.pdf